CLINICAL TRIAL: NCT00415584
Title: Cinacalcet for Treatment of Persistent Secondary Hyperparathyroidism in Renal Transplant Recipients: Effect on Renal Function, Serum Calcium and Bone Histomorphometry
Brief Title: Cinacalcet to Treat Hypercalcemia in Renal Transplant Recipients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Based on information in IRB archives the study was terminated in 2009 due to low enrollment
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Maria Coco, Prof. Dept of Medicine (Nephrology), Montefiore Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-09-244
Record Dates: First submitted 2006-12-21; First posted 2006-12-25 (Estimated); Results first posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Secondary Hyperparathyroidism; Hypercalcemia
Keywords: hypercalcemia; transplant
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Hypercalcemia | interventions — Cinacalcet

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

ARMS (1):
- Cinacalcet Hydrochloride (HCl) (Experimental)
  Interventions: Drug: Cinacalcet HCl

INTERVENTIONS:
Drug: Cinacalcet HCl

SUMMARY:
Secondary hyperparathyroidism can persist following successful renal transplantation and can cause high blood calcium, kidney dysfunction or failure and excessive bone loss among other problems. If the condition does not resolve, surgery is frequently required to remove the parathyroid glands, with all the inherent risks of surgery. Cinacalcet, a medicine used to treat secondary hyperparathyroidism in patients with kidney disease, may be effective in treating this condition in renal transplant recipients. The investigator team will study the effect of cinacalcet on calcium, bone and renal function in a 6 month treatment protocol.

DETAILED DESCRIPTION:
Secondary Hyperparathyroidism in the renal transplant recipient can cause abnormal bone and mineral metabolism, resulting in hypercalcemia that is detrimental to renal function, causing renal dysfunction and calcinosis. These patients often require parathyroidectomy to correct the hypercalcemia. Surgery is not without significant risk to the patient. Risks include vocal cord paralysis, protracted hypocalcemia, cardiac arrhythmias, muscle cramps. In addition, parathyroidectomy has been associated with subsequent renal impairment.

Cinacalcet is a calcimimetic agent that is very effective in the treatment of secondary hyperparathyroidism in patients with renal failure as well as in hypercalcemia of parathyroid cancer. There have been reports of short term Cinacalcet use in renal transplant recipients. Serum calcium was improved in these patients.

However, little is known about the effect of cinacalcet on bone activity and turnover. It is not known whether Cinacalcet causes low turnover bone activity with adynamic bone disease. It is known that low turnover bone disease in renal patients can by itself cause hypercalcemia as the bone becomes static and unable to respond to everyday calcium loads.

Studies have shown that adynamic bone can develop in renal transplant recipients under a variety of conditions. It is not known what effect, if any, cinacalcet has on the bone activity of renal transplant recipients with persistent secondary hyperparathyroidism.

The purpose of the study is to determine the effect of Cinacalcet on serum calcium, renal function and bone histology in renal transplant recipients.

This is a prospective, open-label study. Protocol procedures will include baseline and 6 month measurements of bone mineral density, bone biochemical parameters, glomerular filtration rate, anterior iliac crest bone biopsy. Subjects will start cinacalcet after the first biopsy. The medication will be titrated to normalize serum calcium. Medication will be supplied by the study. Serum electrolytes will be monitored as indicated.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant recipient at least 3 months post transplant
* Hypercalcemic, with serum calcium > 10.5 milliequivalents per liter (mEq/L)
* Persistent hyperparathyroidism, with inappropriately elevated parathyroid hormone (PTH)

Exclusion Criteria:

* Allergic to Cinacalcet HCl, tetracycline
* Pregnant
* On medication that utilizes same liver system as Cinacalcet HCl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-02-09 (Actual); Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Coco, MD, MS, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cinacalcet Hydrochloride (HCl): Cinacalcet Hydrochloride (HCl)
Period: Overall Study
Arm/Group | Cinacalcet Hydrochloride (HCl)
Started | 4
Completed | 3
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Only 4 participants were enrolled into this study.
Groups:
- Cinacalcet HCl: Cinacalcet HCl
Arm/Group | Cinacalcet HCl
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Normalization of Serum Calcium Levels
Description: Serum calcium was to have been assessed by drawing venous blood samples for serum analysis. Normal blood calcium levels for adults range from approximately 8.5 to 10.4 mg/dL, but vary depending on laboratory reference ranges. Changes in serum calcium levels from baseline following treatment with Cinacalcet HCl were to have been summarized and evaluated using paired t-tests.
Time Frame: Baseline to 6 Months
Population: Venous blood samples were not collected and processed and, as such, serum calcium data was not available for this study.
Arm/Group | Cinacalcet HCl
Number analyzed (Participants) | 0

2. Secondary Outcome: Changes in Renal Function
Description: Change in renal function from baseline was to have been assessed at 6 months based on a measurement of Glomerular Filtration Rate (GFR). Normal GFR ranges vary based on age, sex, and body size but are typically > 90 mL/min/1.73 m^2 for healthy individuals. Changes in renal glomerular filtration rate from baseline following treatment with Cinacalcet HCl were to have been summarized and evaluated using paired t-tests.
Time Frame: Baseline to 6 Months
Population: GFR data was not collected for this study and changes in renal function were not able to be assessed.
Arm/Group | Cinacalcet HCl
Number analyzed (Participants) | 0

3. Secondary Outcome: Changes in Bone Mineral Density
Description: Changes in bone mineral density was assessed using central dual energy x-ray absorptiometry (DXA or DEXA). DXA uses radiation to measure how much calcium and other minerals are in a specific area of the bone. For this study, changes in bone mineral density of the left hip, lumbar spine, and left forearm (vs baseline) have been summarized and reported as a percentage change from baseline. Statistical t-tests were not conducted due to limited sample size.
Time Frame: Baseline to 6 Months
Population: Bone mineral density scans taken yielded inconsistent/unreliable results and, as such, powered statistical testing was not conducted. Left forearm scans were only obtained for 3 of the 4 patients.
Measure: Median (Full Range); unit: percentage change from basline
Arm/Group | Cinacalcet HCl
Number analyzed (Participants) | 4
percentage change from basline
  Left Hip | -6.9 [-9.5 to -2.7]
  Spine - Lumbar | -12.9 [-17.3 to -2.4]
  Left Forearm: number analyzed (Participants) | 3
  Left Forearm | -1.2 [-7.1 to -0.6]

4. Other Pre Specified Outcome: Changes in Bone Turnover Rate
Description: Changes in bone turnover rate from baseline were to have been assessed by bone histology and histomorphometry. This was to have been conducted by an examination of bone biopsies, collected after double labeling with tetracycline compounds ~21 days prior to the procedure, to assess for bone turnover and structure. This was to have been a largely observational endpoint as no studies published at the time have described the effect of Cinacalcet HCl on bone histology.
Time Frame: Baseline to 6 Months
Population: Crest bone biopsy samples were collected from the four patients; however, results could not be generalized.
Arm/Group | Cinacalcet HCl
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: Participants were monitored for hospitalizations, infections, rejection episodes, and acute renal failure.
Arm/Group | Cinacalcet HCl
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
Limitations attributable to the collection of DXA bone mineral density scans along with incomplete collections attributable to study design and logistics issues led to incomplete/unreliable results which were unable to be generalized. As indicated in the Change within Bone Mineral Density Outcome Measure, results data for this assessment were limited to basic summaries.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes